CLINICAL TRIAL: NCT03610555
Title: Creating a Patient-centered Report Card for Solid Organ Transplant Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajay Israni, MD (Other)
Responsible Party: Sponsor-Investigator, Ajay Israni, MD, Ajay Israni, M.D., M.S. Nephrologist, Hennepin Healthcare President, Hennepin Healthcare Research Institute, Professor of Medicine Adjunct Faculty School of Public Health, University of Minnesota, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSR#16-4130
Record Dates: First submitted 2018-06-15; First posted 2018-08-01 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Transplants

STUDY DESIGN:
Intervention Model Description: Participants were stratified by transplant center site and block randomized to one of the four groups using permuted block randomization with blocks of size four.
  * Arm 1: SRTR website first, Question 1 first
  * Arm 2: SRTR website first, Question 2 first
  * Arm 3: TCST first, Question 1 first
  * Arm 4: TCST first, Question 2 first
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Other): Sequence 1: SRTR then TCST (Question 1 then Question 2)
  Interventions: Other: Intervention 1 - SRTR (age question 1st)
- Arm 2 (Other): Sequence 2: SRTR then TCST (Question 2 then Question 1)
  Interventions: Other: Intervention 2 - SRTR (BMI question 1st)
- Arm 3 (Other): Sequence 3: TCST then SRTR (Question 1 then Question 2)
  Interventions: Other: Intervention 3 - TCST (age question 1st)
- Arm 4 (Other): Sequence 4: TCST then SRTR (Question 2 then Question 1)
  Interventions: Other: Intervention 4 - TCST (BMI question 1st)

INTERVENTIONS:
Other: Intervention 1 - SRTR (age question 1st) — Participants first viewed the SRTR website to answer Question 1 (Which transplant program within a prespecified area had the most recipients over 70 years of age?). Subsequently, participants crossed over to view the TCST website to answer Question 2 (Which program within a prespecified area had the most recipients with BMI >40?)
  Arms: Arm 1
Other: Intervention 2 - SRTR (BMI question 1st) — Participants first viewed the SRTR website to answer Question 2. Subsequently, participants crossed over to view the TCST website to answer Question 1.
  Arms: Arm 2
Other: Intervention 3 - TCST (age question 1st) — Participants first viewed the TCST website to answer Question 1. Subsequently, participants crossed over to view the SRTR website to answer Question 2.
  Arms: Arm 3
Other: Intervention 4 - TCST (BMI question 1st) — Participants first viewed the TCST website to answer Question 2. Subsequently, participants crossed over to view the SRTR website to answer Question 1.
  Arms: Arm 4

SUMMARY:
Choosing a transplant center that will accept a particular candidate can be difficult and challenging for patients with end-stage organ failure. As transplant centers have varying levels of expertise, interests, and outcomes of solid organ transplant, patient health-related characteristics influence the variation in candidates centers will accept. Most transplant candidates undergo waitlist work-ups as outpatients and many undergo transplant at centers not closest to their homes. Some are listed at more than one center. Several studies suggest that patients have a choice of centers. The PI, as Deputy Director of the Scientific Registry of Transplant Recipients (SRTR), provides comparative information to the public about each solid organ transplant center in the United States. The risk adjusted outcomes, in the report cards, account for the transplant recipient's health-related characteristics, donor characteristics and transplant related factors. Unfortunately, in their current format, the report cards are not designed for transplant candidates, many of whom may have low health literacy and numeracy.

The proposed work aims to develop and evaluate a patient-centered website and printouts of the SRTR report cards that will effectively communicate comparative information to transplant candidates about their alternatives when choosing transplant centers. We will develop a novel tool to allow candidates to tailor the report cards to their clinical profiles based on their health-related characteristics and to communicate information on alternative transplant centers that perform transplants in patients like them. Aim 1 will use focus groups to determine which transplant center characteristics to present to transplant candidates and how to present these characteristics clearly in a patient centered report card. Using this information, Aim 2 will develop a patient-centered website and printouts of the SRTR report card that effectively communicate comparative information about transplant centers to transplant candidates. Lastly, Aim 3 will conduct a randomized clinical trial to evaluate the effectiveness of the patient centered SRTR report card. We will determine transplant candidates' comprehension and the value of the comparative quality reports, and the effect on clinical decision making and status on the waiting list. After the RCT, a convenience sample of online visitors to the new website will be assessed for similar outcomes.

DETAILED DESCRIPTION:
Before the intervention, the study design with use of hypothetical scenarios will be explained to the participant. The concept of randomization will be also be explained. The participants will be asked a few questions to assess their understanding of the study design, specifically the hypothetical nature of the scenarios. We will also assess whether they understand the concept of being randomized to see one website first and then the other. Only those participants that understand the study design will be invited to participate in the intervention and will be randomized. For subjects that are randomized, a survey will be administered verbally to collect demographic information and information about their kidney disease and comorbidities. The functional health literacy and numeracy assessment and health status questionnaire will be completed. Subjects will be stratified by the transplant center site and then block randomized. One group will be shown the existing SRTR website with its existing SRTR report cards and then the website with the new patient-centered AHRQ report cards for kidney transplants. The other group will be shown the two websites in opposite order. Each participant will have at most 30 minutes to view each of the websites. After viewing each website, responses to the intervention will be collected. Sessions where participants are reviewing the websites will be recorded using Zoom. Figure 2 shows the study design whereby subjects will be block randomized once to one of the four groups consisting of 18 subjects each. At the end of the study, the patients will have access to both the websites.

The study interventions can be administered in person on a laptop. During the COVID-19 pandemic, the intervention can be administered remotely via email and zoom. The link to the websites will be sent via encrypted email and the intervention will be recorded via zoom. The recordings for subjects at Hennepin Healthcare will be stored on computers at that site.

If participant does not have your own electronic device or internet, the study will send the participant a study iPad with internet that participant can use for the intervention and then to send back to the study team. We will provide detailed instructions on how to use the iPad and Zoom application. The study will also pay for a FedEx pick up from the participants' home to return the iPad to the study team after the completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

All adults seeking a kidney transplant are eligible for the RCT. We will focus on recruiting kidney waitlist candidates.

Exclusion criteria:

are inability to speak or understand English, visual impairment, and inability to give consent. All vulnerable populations except for those listed in the table titled vulnerable populations, will be excluded.

.

.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HCMC, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Israni AK, Schladt D, Bruin MJ, Chu S, Snyder JJ, Hertz M, Valapour M, Kasiske B, McKinney WT, Schaffhausen CR. Deconstructing Silos of Knowledge Around Lung Transplantation to Support Patients: A Patient-specific Search of Scientific Registry of Transplant Recipients Data. Transplantation. 2022 Aug 1;106(8):1517-1519. doi: 10.1097/TP.0000000000004051. Epub 2022 Feb 11. No abstract available. PMID 35152256
- [Background] Chu S, Bruin MJ, McKinney WT, Israni AK, Schaffhausen CR. Design of a patient-centered decision support tool when selecting an organ transplant center. PLoS One. 2021 May 17;16(5):e0251102. doi: 10.1371/journal.pone.0251102. eCollection 2021. PMID 33999964
- [Background] McKinney WT, Schaffhausen CR, Schladt D, Bruin MJ, Chu S, Snyder JJ, Martin C, Alexy T, Kasiske B, Israni AK. Designing a patient-specific search of transplant program performance and outcomes: Feedback from heart transplant candidates and recipients. Clin Transplant. 2021 Feb;35(2):e14183. doi: 10.1111/ctr.14183. Epub 2020 Dec 19. PMID 33617066
- [Background] McKinney WT, Schaffhausen CR, Bruin MJ, Chu S, Schladt D, Matas A, Snyder J, Kasiske B, Israni AK. Development of a Patient-specific Search of Transplant Program Outcomes and Characteristics: Feedback From Kidney Transplant Patients. Transplant Direct. 2020 Jul 17;6(8):e585. doi: 10.1097/TXD.0000000000001036. eCollection 2020 Aug. PMID 32766433
- [Background] Schaffhausen CR, Bruin MJ, McKinney WT, Snyder JJ, Matas AJ, Kasiske BL, Israni AK. How patients choose kidney transplant centers: A qualitative study of patient experiences. Clin Transplant. 2019 May;33(5):e13523. doi: 10.1111/ctr.13523. Epub 2019 Apr 21. PMID 30861199
- [Background] Schaffhausen CR, Bruin MJ, Chu S, Wey A, McKinney WT, Snyder JJ, Lake JR, Matas AJ, Kasiske BL, Israni AK. Comparing Pretransplant and Posttransplant Outcomes When Choosing a Transplant Center: Focus Groups and a Randomized Survey. Transplantation. 2020 Jan;104(1):201-210. doi: 10.1097/TP.0000000000002809. PMID 31283676
- [Result] McKinney WT, Israni K, Schaffhausen CR, Schladt DP, Lyden GR, Matas A, Wolf J, Japuntich S, Israni AK. Randomized Controlled Trial to Evaluate a New Tool to Support Patient Decision-making on Transplant Centers. Clin Transplant. 2024 Dec;38(12):e70043. doi: 10.1111/ctr.70043. PMID 39620865
- See also: This website is the finalized version of the intervention study site. — https://transplantcentersearch.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults (age 18+) were recruited to participate from the waiting list or in the process of being evaluated for deceased donor kidney transplants at two urban transplant programs in the Midwest. Patients were approached by mail with follow-up via a phone call with an institutional review board-approved script for attaining consent and conducting the intervention.
Pre-assignment Details: A total of (n=6) were excluded from the study. Reasons for exclusion include the following: Not meeting exclusion criteria (n=1) and excluded since part of vanguard study (n=5).
Groups:
- Arm 1: Sequence1: Participants first viewed the SRTR website to answer Question 1 (Which transplant program within a prespecified area had the most recipients over 70 years of age?). Subsequently, participants crossed over to view the TCST website to answer Question 2 (Which program within a prespecified area had the most recipients with BMI >40?).
- Arm 2: Sequence2: Participants first viewed the SRTR website to answer Question 2. Subsequently, participants crossed over to view the TCST website to answer Question 1.
- Arm 3: Sequence3: Participants first viewed the TCST website to answer Question 1. Subsequently, participants crossed over to view the SRTR website to answer Question 2.
- Arm 4: Sequence4: Participants first viewed the TCST website to answer Question 2. Subsequently, participants crossed over to view the SRTR website to answer Question 1.
Period: Initial Randomization
Arm/Group | Arm 1: Sequence1 | Arm 2: Sequence2 | Arm 3: Sequence3 | Arm 4: Sequence4
Started | 12 | 19 | 18 | 19
Completed | 12 | 19 | 18 | 19
Not Completed | 0 | 0 | 0 | 0
Period: Crossover to 2nd Website and Question
Arm/Group | Arm 1: Sequence1 | Arm 2: Sequence2 | Arm 3: Sequence3 | Arm 4: Sequence4
Started | 12 | 19 | 18 | 19
Completed | 12 | 18 | 17 | 19
Not Completed | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: SRTR Website First, Question 1 First: Show patient SRTRT website first, then question 1 first
- Arm 2: SRTR Website First, Question 2 First: Show patient SRTRT website first, then question 2 first
- Arm 3: TCST First, Question 1 First: Show patient TCST website first, then question 1 first.
- Arm 4: TCST First, Question 2 First: Show patient TCST website first, then question 2 first.
- Total: Total of all reporting groups
Arm/Group | Arm 1: SRTR Website First, Question 1 First | Arm 2: SRTR Website First, Question 2 First | Arm 3: TCST First, Question 1 First | Arm 4: TCST First, Question 2 First | Total
Number analyzed (Participants) | 12 | 19 | 18 | 19 | 68
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 9 | 6 | 28
  Male | 7 | 11 | 9 | 13 | 40
Education Level [Count of Participants; unit: Participants] — Captures educational attainment
  Participants
    Less than high school | 0 | 1 | 1 | 0 | 2
    High School | 2 | 8 | 3 | 2 | 15
    Some college | 4 | 2 | 8 | 4 | 18
    More than college (e.g. M.A., PHD, MD) | 1 | 4 | 5 | 7 | 17
    College | 5 | 4 | 1 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-Hispanic White | 9 | 11 | 12 | 17 | 49
  Race: African American | 3 | 5 | 4 | 2 | 14
  Race: Other | 0 | 3 | 2 | 0 | 5
Single Item Literacy Scale (score >2) [Count of Participants; unit: Participants] — Evaluates subjective literacy; scores > 2 indicate need for assistance when reading health related materials
  Participants
    Yes | 0 | 6 | 3 | 2 | 11
    No | 12 | 13 | 15 | 17 | 57
Single Item Literacy Scale (mean) [Mean (Standard Deviation); unit: Score on a scale] — Evaluate mean scores on Single Item Literacy Scale; scores range from 1 - 5. Scores greater than 2 indicate some difficulty with health literacy.
  Score on a scale | 1.33 (0.49) | 1.84 (1.01) | 1.39 (0.78) | 1.47 (0.84) | 1.53 (0.84)
Age, Customized [Count of Participants; unit: Participants]
  Age: <50 years | 1 | 4 | 3 | 6 | 14
  Age: 50 < 65 years | 3 | 10 | 10 | 8 | 31
  Age: 65+ years | 7 | 5 | 5 | 5 | 22
  Age: Missing | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Ethnicity: Latino | 0 | 1 | 1 | 3 | 5
    Ethnicity: Non-Latino | 12 | 18 | 17 | 15 | 62
    Ethnicity: Missing | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Correct Response to Question 1 and 2
Description: The primary outcome is the comprehension of the report card. To assess comprehension, the correct response to the following question will be assessed, "Which transplant program within a prespecified area had the most recipients over 70 years of age; and which programs had the most recipients with BMI >40"
Time Frame: 30 minutes
Population: To assess comprehension, the correct response to the following question will be assessed, "Which transplant program within a prespecified area had the most recipients over 70 years of age; and which programs had the most recipients with BMI >40"
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: SRTR Website First, Question 1 First | Arm 2: SRTR Website First, Question 2 First | Arm 3: TCST First, Question 1 First | Arm 4: TCST First, Question 2 First
Number analyzed (Participants) | 12 | 18 | 18 | 19
Participants
  Comprehension : Question 1 - age over 70 | 5 | 17 | 17 | 11
  Comprehension : Question 2 - BMI | 12 | 17 | 16 | 18
  Missing : Question 1 - age over 70 | 0 | 0 | 0 | 0
  Missing : Question 2 - BMI | 0 | 0 | 1 | 0

2. Secondary Outcome: Perceived Value of Information
Description: Perceived value of information will be determined via patient responses to the following question, "How useful is the information in the report card in helping you choose a transplant center for you or your family?" Response choices to the questions will be based on a 5-point Likert-type scale (1 = extremely useful to 5 = not useful at all; score 1 indicates the better outcome and score 5 indicates worse outcome).
Time Frame: 30 minutes
Population: 1 participant did not respond to the study question and 1 participant was unable to view the Current website. Using an intention to treat approach, we included both participants in the final analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Current Website: Show patient one of the website
- New Patient Centered Website: Show patient another (different) of the website
  new patient centered website
Arm/Group | Current Website | New Patient Centered Website
Number analyzed (Participants) | 68 | 68
units on a scale | 2.16 (1.03) | 1.97 (1.02)

3. Secondary Outcome: Measurement of Satisfaction With Decision Making
Description: We measured satisfaction with decision-making and decisional conflict using the Ottawa Decisional Conflict Scale (DCS). Participants were asked to answer four items to assess satisfaction with decision making. These four items are: a) summed; b) divided by 4; and c) multiplied by 25. Scores ranges from 0 [great satisfaction] to 100 [lower satisfaction].
Time Frame: 30 minutes
Population: This was a cross-over study design.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Current Website | New Patient Centered Website
Number analyzed (Participants) | 68 | 68
units on a scale | 15.5 (19.6) | 13.4 (19.7)

ADVERSE EVENTS:
Time Frame: Throughout the study session (approximately 1.5 hours).
Description: Adverse events were monitored via non-systematic assessment (researcher observation) during the 1.5-hour study session.
Groups:
- Current Website: Show patient one of the websites.
  The risks for participating in the study are not higher than a conversation they have in their daily life. They were shown a website and responded a few questions.
- New Patient Centered Website: Show patient another (different) of the website
  The risks for participating in the study are not higher than a conversation they have in their daily life. They were shown a website and responded a few questions.
Arm/Group | Current Website | New Patient Centered Website
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/68 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT03610555/Prot_SAP_000.pdf